CLINICAL TRIAL: NCT00405964
Title: Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter/Multinational, Efficacy and Safety Study of Desloratadine 5 mg in the Treatment of Subjects With Allergic Rhinitis Who Meet the Criteria for Persistent Allergic Rhinitis (PER)
Brief Title: Study for the Treatment of Persistent Allergic Rhinitis With Desloratadine (Study P04684)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04684
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-mg Desloratadine tablet (Experimental)
  Interventions: Drug: 5-mg Desloratadine
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 5-mg Desloratadine — 5-mg Desloratadine tablet, once daily for 12 weeks
  Other Names: SCH 34117, Aerius
  Arms: 5-mg Desloratadine tablet
Drug: Placebo tablet — Placebo tablet, once daily for 12 weeks
  Arms: Placebo tablet

SUMMARY:
This study will investigate the effectiveness of desloratadine in treating subjects with allergic rhinitis who meet the criteria for persistent allergic rhinitis (PER)

ELIGIBILITY:
Inclusion Criteria:

* For this study, the diagnosis of persistent allergic rhinitis (PER) is not based solely on the current episode of allergic rhinitis (AR). Subjects must have at least a 2 year history of AR consistent with PER (defined as symptoms of allergic rhinitis present more than four days per week and for more than four consecutive weeks per year); the current episode can count as the second year.
* Subjects must be 12 years of age and older, of either sex and of any race.
* At the Run-in Visit, subjects must be sufficiently symptomatic, with a T5SS 12-hour AM-PRIOR (Subject's Status Over Previous 12 Hours) symptoms severity score of at least 8.
* In order for a subject to qualify at the Baseline Visit, the sum of the daily averages of the diary recordings of the 12-hour AM PRIOR + PM-PRIOR T5SS collected during Days -4 to -1 and the AM PRIOR T5SS on the morning of the Baseline Visit (Day 1) must be >=40.
* Subjects must have a positive skin-prick test at screening to one or more allergens in the Global Allergy and Asthma European Network (GA2LEN) (or the usually used local) panel of seasonal and perennial allergens. Subjects must demonstrate an antigen-induced skin prick wheal at least 3 mm in diameter greater than diluent control. The positive tests must include the allergen(s) prevalent while this study is active.
* Subjects must be free of any clinically significant disease, other than PER, which would interfere with the study evaluations.
* Subjects, or parents or legal guardians, must give written informed consent. Subjects must be able to adhere to dose, visit schedules and meet study requirements.
* In females of childbearing potential, the urine pregnancy test (human chorionic gonadotropin [hCG]) must be negative at the Screening Visit.
* Nonsterile or premenopausal female subjects must be using a medically accepted method of birth control, that is, oral contraceptive, hormonal implant, medically prescribed intra-uterine device (IUD), or depot injectable during the entire study. A female subject who is not currently sexually active must agree and consent to use one of the above-mentioned methods, if she becomes sexually active while participating in the study. A female subject who is not of childbearing potential must have a medical record of being surgically sterile (for example, hysterectomy, and tubal ligation), or be at least 1 year postmenopausal.

Exclusion Criteria:

* Subjects with a history of anaphylaxis and/or severe local reactions(s) to skin testing with allergens.
* Subjects with intolerable symptoms that would make participating in the study unbearable.
* Subjects who have had an upper respiratory tract or sinus infection that required antibiotic therapy, and have not had at least a 14-day washout prior to the run-in period, or who have had a viral upper respiratory infection within 7 days prior to screening.
* Subjects with asthma who require chronic use of inhaled or systemic corticosteroids.
* Subjects with a current history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* Subjects on immunotherapy (desensitization therapy) unless on a regular maintenance schedule prior to Visit 1 and staying on this schedule for the remainder of the study.
* Subjects who, in the opinion of the investigator, are dependent on nasal, oral or ocular decongestants, nasal topical antihistamines or nasal steroids.
* Subjects who have used any drug or device in an investigational protocol in the 30 days prior to Visit 1.
* Female subjects who are pregnant or nursing.
* Subjects with a history of hypersensitivity to the study drug or to their excipients or known to not tolerate any antihistamine.
* Subject is a member of the Investigational Study Staff (currently involved with this study) or a member of the staff's family.
* Subjects with current evidence of clinically significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune disease, or other disease that preclude the subject's participation in the study.
* Subjects whose ability to provide informed consent is compromised.
* Subjects with a history of noncompliance with medications or treatment protocols.
* Subjects with rhinitis medicamentosa.
* Subjects who have, in the opinion of the investigator or designee, clinically significant nasal structural abnormalities, including large nasal polyps or marked septum deviation, that significantly interferes with nasal air flow.
* Subjects who have not observed mediation washout times prior to visit 2

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bousquet J, Bachert C, Canonica GW, Mullol J, Van Cauwenberge P, Jensen CB, Fokkens WJ, Ring J, Keith P, Gopalan G, Lorber R, Zuberbier T; ACCEPT-2 Study Group. Efficacy of desloratadine in persistent allergic rhinitis - a GA(2)LEN study. Int Arch Allergy Immunol. 2010;153(4):395-402. doi: 10.1159/000316351. Epub 2010 Jun 18. PMID 20559006
- [Derived] Bousquet J, Zuberbier T, Canonica GW, Fokkens WJ, Gopalan G, Shekar T. Randomized controlled trial of desloratadine for persistent allergic rhinitis: correlations between symptom improvement and quality of life. Allergy Asthma Proc. 2013 May-Jun;34(3):274-82. doi: 10.2500/aap.2013.34.3668. PMID 23676577

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-mg Desloratadine Tablet: Desloratadine 5 mg orally daily. Dosing was to be in the morning (AM) within 1 hour of awakening.
- Placebo Tablet: Matching placebo, orally daily.
Period: Overall Study
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Started | 360 | 356
Completed | 301 | 261
Not Completed | 59 | 95
Not completed — Treatment Failure | 17 | 45
Not completed — Adverse Event | 7 | 16
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 19 | 23
Not completed — Protocol Violation | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet | Total
Number analyzed (Participants) | 360 | 356 | 716
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 348 | 341 | 689
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (12.1) | 33.9 (12.3) | 33.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 198 | 406
  Male | 152 | 158 | 310

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant's AM/PM PRIOR Total 5 Symptom Score (T5SS) Over Days 1 to 29 of Treatment
Description: AM/PM PRIOR (the participant's status over previous 12 hours) T5SS from the participant's daily diary averaged over treatment Days 1 to 29. AM/PM is the average of separate morning (AM) and evening (PM) evaluations. Scores were defined for T5SS as 0: no symptoms to 15: all severe symptoms. A two-way analysis of variance (ANOVA) model with treatment and site effects was used to examine the treatment difference.
Time Frame: Baseline and Days 1-29
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 355 | 351
units on a scale
  Baseline | 9.63 (0.13) | 9.55 (0.12)
  Days 1-29 | -3.76 (0.22) | -2.87 (0.21)
Statistical Analysis 1: Comparison: 5-mg Desloratadine Tablet vs Placebo Tablet; Test type: Superiority or Other; p < .001, ANOVA — Determined for site. P-value of <.001 for treatment as well

2. Secondary Outcome: Change From Baseline in the Total Rhinoconjunctivitis Quality of Life Questionnaire-Standarized Version (RQLQ-S) After 29 Days of Treatment
Description: The RQLQ-S was only completed for participants above 18 years of age. The RQLQ-S was not available for participants 12 to 17 years of age. This questionnaire asked questions pertaining to daily activities, sleep, non-nose eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotions. The scale went from 0 (not troubled) to 6 (extremely troubled). A two-way analysis of variance (ANOVA) model with treatment and site effects was used to examine the treatment difference.
Time Frame: Baseline and Day 29
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 313 | 289
units on a scale
  Baseline | 3.30 (0.08) | 3.15 (0.08)
  Day 29 | -1.35 (0.10) | -0.95 (0.10)
Statistical Analysis 1: Comparison: 5-mg Desloratadine Tablet vs Placebo Tablet; Test type: Superiority or Other; p = 0.035, ANOVA — Determined for site. Treatment p-value <.001

3. Secondary Outcome: Change From Baseline in Participant's AM/PM PRIOR T5SS Over Days 1 to 85 of Treatment
Description: AM/PM PRIOR (the participant's status over previous 12 hours) T5SS from the participant's daily diary averaged over treatment Days 1 to 85. AM/PM is the average of separate AM and PM evaluations. Scores were defined for T5SS as 0: no symptoms to 15: all severe symptoms. A two-way analysis of variance (ANOVA) model with treatment and site effects was used to examine the treatment difference.
Time Frame: Baseline and Days 1-85
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 355 | 351
units on a scale
  Baseline | 9.63 (0.13) | 9.55 (0.12)
  Days 1-85 | -4.50 (0.23) | -3.61 (0.23)
Statistical Analysis 1: Comparison: 5-mg Desloratadine Tablet vs Placebo Tablet; Test type: Superiority or Other; p < .001, ANOVA — Same p-value for treatment and site

ADVERSE EVENTS:
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 1/360 | 2/356
Other Adverse Events (participants affected / at risk) | 60/360 | 48/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-mg Desloratadine Tablet (N=360) | Placebo Tablet (N=356)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-mg Desloratadine Tablet (N=360) | Placebo Tablet (N=356)
Nasopharyngitis (Infections and infestations) | 38 (44) | 17 (18)
Headache (Nervous system disorders) | 25 (45) | 37 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less